CLINICAL TRIAL: NCT01562223
Title: Repeatability Assessment of Quantitative DCE-MRI and DWI: A Multicenter Study of Functional Imaging Standardization in the Prostate
Brief Title: Studying Repeated DCE-MRI and DWI in Patients Diagnosed With Prostate Cancer
Acronym: A6701QIBA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000728901; ACRIN-6701 (Other: ACRIN Foundation); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2012-03-22; First posted 2012-03-23 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: stage IIA prostate cancer; stage IIB prostate cancer; stage III prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — motexafin gadolinium; Gadolinium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Repeatability Assessment (Experimental): Gadolinium motexafin gadolinium All participants will undergo two consecutive DCE-MRI and DWI scans per same imaging parameters and subsequent comparison for repeatability.
  Interventions: Other: motexafin gadolinium

INTERVENTIONS:
Other: motexafin gadolinium
  Other Names: Gadolinium

SUMMARY:
RATIONALE: Diagnostic procedures, such as dynamic contrast-enhanced magnetic resonance imaging or DCE-MRI and diffusion-weighted imaging or DWI, may provide images of prostate cancer or any cancer that remains after biopsy.

PURPOSE: This trial studies repeated DCE-MRI and DWI in patients diagnosed with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the test-retest performance, assessed by the repeatability coefficient [RC] of K^trans and gadolinium curve (IAUGC90^bn) and measured by median pixel values of the whole prostate.
* Determine the test-retest performance, assessed by the RC of diffusion-weighted imaging (DWI) metrics D(t) and measured by median pixel values of the whole prostate.

Secondary

* Determine the test-retest performance, assessed by RC of K^trans, IAUGC90^bn, and D(t), and measured by median pixel values of the dominant prostate tumor.
* Determine the effect of reader on the RC of dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI) and DWI metrics for whole prostate and tumor nodule target lesion.
* Determine whether T1-dependent or T1-independent methods for gadolinium quantification in DCE-MRI studies produce differing values for the RC for K^trans and IAUGC90^bn.
* Explore the correlation between DCE-MRI and DWI metrics for both whole prostate and dominant tumor nodule as target lesions. (Exploratory)
* Determine whether the "coffee break" approach toward test-retest analysis of quantitative DWI provides a reasonable estimate of the RC of D(t)of the whole prostate, using as the gold standard the RC of D(t) obtained between the two separate MRI visits. (Exploratory)

OUTLINE: This is a multicenter study. Patients are stratified according to MRI vendor used (Siemens vs GE vs Philips).

Patients receive gadolinium-based contrast IV and undergo DCE-MRI* and DWI 2 imaging at 2-14 days apart prior to treatment initiation. A central reader evaluation of the 2 successive scans is then conducted.

NOTE: *At the discretion of the participating sites, the initial MRI visit (MRI SCAN 1) may be supplemented with endorectal-coil imaging per institutional norms.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of prostate adenocarcinoma by transrectal ultrasound (TRUS)-guided biopsy between 28 to 90 days prior to enrollment
* Minimal tumor burden as defined by at least one of the following criteria:

  * One single core with ≥ 50% cancer burden and ≥ 5 mm tumor length
  * Two or more cores in the same prostate region, each with ≥ 30% cancer burden
  * Three or more cores positive for prostate cancer (of any magnitude of cancer burden) in the same prostate region
  * Gleason score of 7 or higher cancer burden
  * Prostate-specific antigen (PSA) ≥ 10 ng/mL

PATIENT CHARACTERISTICS:

* Able to tolerate magnetic resonance imaging (MRI) required by protocol, to be performed at an American College of Radiology Imaging Network (ACRIN)-qualified facility and scanner
* Not suitable to undergo MRI or gadolinium-based contrast agent because of:

  * Severe claustrophobia not relieved by oral anxiolytics per institutional standard practice
  * Presence of MRI-incompatible metallic objects or implanted medical devices in body (including, but not limited to, non-MRI compatible metal objects, cardiac pacemaker, aneurysm clips, artificial heart valves with steel parts, or metal fragments in the eye or central nervous system)
  * Renal failure, as determined by glomerular filtration rate (GFR) < 30 mL/min based on a serum creatinine level obtained within 48 hours prior to enrollment
  * Weight greater than that allowable by the MRI table, per local institutional practice

PRIOR CONCURRENT THERAPY:

* No anti-androgenic therapy within 30 days prior to enrollment
* No prior external-beam radiotherapy, proton radiotherapy, or brachytherapy to the prostate
* No prior hip replacement or other major pelvic surgery

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08-27 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Repeatability assessment of DCE-MRI metrics Ktrans and blood-normalized initial area under the gadolinium curve (IAUGC90bn) and the DWI metric D(t) | 2 to 14 Days
  The repeatability coefficient (RC) and its 95% confidence interval (CI) will be estimated for each metric [ ktrans, IAUGC90bn] using the method of Barnhart and Barboriak, 2009

SECONDARY OUTCOMES:
Test-retest performance, assessed by the RC of Ktrans, IAUGC90bn, and D(t), and measured by median pixel values of the prostate tumor | 2 to 14 Days
  The repeatability coefficient (RC) and its 95% confidence interval (CI) will be estimated for each metric using the method of Barnhart and Barboriak, 2009
Comparison between T1-dependent or T1-independent methods for gadolinium quantification produce differing values for the RC for Ktrans | 2 to 14 Days
  The repeatability coefficient (RC) and its 95% confidence interval (CI) will be estimated for each metric ktrans] and each method [ independent and dependent] using the method of Barnhart and Barboriak, 2009

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Rosen, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
See ACRIN data Sharing Policy:
  https://www.acrin.org/RESEARCHERS/POLICIES/DATAANDIMAGESHARINGPOLICY.aspx

REFERENCES:
- See also: National Cancer Institute's clinical trials database — https://clinicaltrials.gov/ct2/show/NCT01562223